CLINICAL TRIAL: NCT03608046
Title: Avelumab Combined With Cetuximab and Irinotecan for Treatment Refractory Metastatic Colorectal Microsatellite Stable Cancer - A Proof of Concept, Open Label Non-randomized Phase IIa Study. The AVETUXIRI Trial
Brief Title: Avelumab Combined With Cetuximab and Irinotecan for Treatment Refractory Metastatic Colorectal Microsatellite Stable Cancer
Acronym: AVETUXIRI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL-mCRC-2018-MS100070-0095
Record Dates: First submitted 2018-07-16; First posted 2018-07-31 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Colorectal Neoplasms, Malignant
MeSH Terms: conditions — Colonic Neoplasms | interventions — avelumab; Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab, Cetuximab, Irinotecan (Experimental): Avelumab : administrated at a fixed dose of 10 mg/kg once every 2- week. Cetuximab: administered at 400 mg/m2 loading dose week 1, 250 mg/m2 from week 2 followed by 500 mg/m2 from week 3.
  Irinotecan: administrated every 2 weeks (180 mg/m2).
  Interventions: Drug: Avelumab; Drug: Cetuximab Injection; Drug: Irinotecan

INTERVENTIONS:
Drug: Avelumab — Avelumab will be administered at a fixed dose of 10 mg/kg once every 2- week
Drug: Cetuximab Injection — Cetuximab will be administered at 400 mg/m2 loading dose week 1, 250 mg/m2 from week 2 followed by 500 mg/m2 from week 3 and irinotecan administered every 2 weeks (180 mg/m2).
Drug: Irinotecan — Irinotecan will be administered every 2 weeks (180 mg/m2)

SUMMARY:
Cancer immunotherapy with immunostimulatory antibodies targeting the CTLA-4 or PD-1/PD-L1 pathways has demonstrated its efficacy in variable proportions of cancer. For metastatic colorectal cancer (mCRC) it appeared that only the small subgroup of patients with MSI-H tumors (microsatellite instability-high phenotype) had a clinically meaningful response to the anti-PD-1- L1 antibodies. In the majority group of non-MSI-H CRC (90-95% of patients), current research expect that additional means would be able to render the tumor "immunogenic" (like MSI-H CRC) and increase the intratumoral immune infiltrate which is the prerequisite to observe a benefit from PD1-PD-L1 inhibitors. Combinations of immune checkpoint inhibitors and procedures that increase intratumoral immune responses, such as targeted therapy, are actively explored.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over, Performance status: ECOG 0-1
* Histologically proven metastatic colorectal adenocarcinoma, refractory to standard chemotherapy (fluoropyrimidine, oxaliplatin, irinotecan) and anti-EGFR treatment (only for RAS WT tumor)
* Measurable disease (RECIST 1.1)
* Metastasis accessible for sequential biopsies
* Patient consent for metastasis biopsies in the study protocol
* BRAF V600E wild-type and MSS tumors
* Adequate normal organ and marrow function (see adequate section of the full protocol for definition)
* Life expectancy of at least 4 months

Exclusion Criteria:

* Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy that are not indicated in the study protocol
* Systemic autoimmune disease,
* Chronic treatment with corticoids or other immunosuppressive treatment
* Clinically significant cardiac, lung or general disease despite optimal treatment
* Non-progressive disease following irinotecan-based treatment.
* For RAS WT, non-progressive disease following anti-EGFR treatment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2018-10-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate | Up to 19 weeks
  The overall tumor response rate (ORR) defined as the proportion of all included patient with a confirmed best overall tumor response of PR or CR according to irRECIST 1.1 occuring until 19 weeks after study treatment start.

SECONDARY OUTCOMES:
Adverse events | Up to 19 weeks
  Safety will be controlled

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi

REFERENCES:
- [Derived] Huyghe N, Benidovskaya E, Masoodi T, Sinapi I, De Cuyper A, Vempalli F, Beyaert S, Bouzin C, Osorio FM, Ferraro L, van Baren N, Helaers R, Goffette P, Ghaye B, van Maanen A, Castella ML, Ceccarelli M, Bedognetti D, Galon J, Hendrickx WRL, Carrasco J, Van den Eynde M. Impact of the tumor immune contexture in microsatellite-stable metastatic colorectal cancer treated with avelumab, cetuximab, and irinotecan. Cell Rep Med. 2025 Jul 15;6(7):102201. doi: 10.1016/j.xcrm.2025.102201. Epub 2025 Jun 24. PMID 40562041